CLINICAL TRIAL: NCT06549387
Title: Topo-Pachymetric Customized Accelerated Epithelium-On Versus Standard Accelerated Epithelium-Off Corneal Collagen Cross Linking in the Management of Keratoconus
Brief Title: Topo-Pachymetric Customized Accelerated Epi-On Vs Accelerated Epi-Off Corneal Cross Linking in Keratoconus Management
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Paula Sameh Youssef, M.Sc., Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: _MD-402-2023_
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Amount of Corneal Flattening (Kmax Flattening); Change in the Endothelial Cell Count
MeSH Terms: interventions — Corneal Cross-Linking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The topo-pachimetric customized accelerated epithelium-On (aCFXL group) (Active Comparator)
  Interventions: Procedure: Corneal cross linking
- The standard accelerated CXL (aCXL) protoco (Active Comparator)
  Interventions: Procedure: Corneal cross linking
- Progressive Fluence Epi-on accelerated crosslinking M nomogram (Active Comparator)
  Interventions: Procedure: Corneal cross linking

INTERVENTIONS:
Procedure: Corneal cross linking — Applying UVA irradiation to the cornea after soaking with riboflavin

SUMMARY:
The objective of this study is to compare the clinical effectiveness and safety of Topo-Pachymetric Customized Accelerated Epithelium-On (aCFXL) to Standard Accelerated Epithelium-Off (aCXL) Corneal Collagen Cross-Linking in the management of keratoconus. The study aims to evaluate visual and structural outcomes, to provide valuable insights into optimizing treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years or older
2. Corrected distance visual acuity (CDVA) of ≥ 0.3 Snellen.
3. Central corneal thickness (de-epithelialized) of ≥ 400 micron.
4. Corneal endothelial count of ≥ 2000.

Exclusion Criteria:

1. Previous eye surgery
2. The presence of lesions other than keratoconus, central or paracentral scaring
3. History of Cross linking
4. History of viral keratitis
5. Connective tissue diseases
6. Pregnancy or lactation during the study.
7. The presence of nystagmus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Amount of corneal flattening | 6 months
  Kmax flattening
Change in the endothelial cell count. | 6 months
  the stability or decrease in the endothelial cell count.

SECONDARY OUTCOMES:
Best corrected visual acuity | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al Ainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided